CLINICAL TRIAL: NCT02101255
Title: Effect of Curodont™ Repair in Patients With Early Approximal Carious Lesions: A Mono-centre, Controlled, Single-blinded, Randomised, Split-mouth, Post-marketing Study
Brief Title: Effect of Curodont™ Repair in Patients With Early Approximal Carious Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Credentis AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P11-4-RACL
Record Dates: First submitted 2014-03-21; First posted 2014-04-02 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Dental Caries
Keywords: Dental caries; Curodont Repair; P11-4
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curodont Repair (Experimental): Application on Day 0 and Day 360
  Interventions: Device: Curodont Repair
- Fluoride (Active Comparator): Application on Day 0, Day 180, Day 360, Day 540
  Interventions: Device: Fluoride

INTERVENTIONS:
Device: Curodont Repair — Self-assembling peptide, biomimetic re-mineralisation
  Application on Day 0 and Day 360
  Other Names: P11-4
  Arms: Curodont Repair
Device: Fluoride — Application on Day 0, Day 180, Day 360, Day 540
  Other Names: Duraphat
  Arms: Fluoride

SUMMARY:
The purpose of this study is to evaluate the therapeutic benefit of Curodont Repair for the treatment of early approximal carious lesions compared to fluoride.

DETAILED DESCRIPTION:
All study participants must have two early approximal carious lesions in need of a treatment but not of an invasive treatment (split-mouth design). One lesion will be treated with Curodont Repair and one with fluoride as control. Study duration is 24 months. For assessment x-ray pictures, Diagnodent Pen and DiagnoCam is used.

ELIGIBILITY:
Inclusion Criteria:

1. Two approximal carious lesions on different teeth with at least one tooth in between
2. Both study lesions must not require an invasive treatment
3. Size and form of the lesions: the lesions must be fully visible and assessable on radiographs
4. The two carious lesions must fall into classes:

   * D2 (inner half of enamel)
   * D3 (outer part of dentine) but only if very little dentine is involved (enamel-dentine junction)
5. Able and willing to observe good oral hygiene throughout the study
6. Age ≥ 18 years and ≤ 65 years
7. Willing and able to attend the on-study visits
8. Willing and able to understand all study-related procedures
9. Written informed consent before participation in the study

Exclusion Criteria:

1. The two study test lesions are located on adjacent teeth
2. Fluoride varnish application < 3 months prior to study treatment
3. Tooth with numerous carious lesions
4. Evidence of tooth erosion
5. History of head and neck illnesses (e.g. head/neck cancer)
6. Any pathology or concomitant medication affecting salivary flow or dry mouth
7. Any metabolic disorders affecting bone turnover
8. Patient suffers from diabetes
9. Concurrent participation in another clinical trial
10. Women who are breast-feeding, pregnant or who plan a pregnancy during the study
11. Women of childbearing potential who declare being unwilling or unable to practice contraception such as hormonal contraceptives, sexual abstinence or intercourse with a vasectomised partner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-07; Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Opaqueness on X-Ray | Day 360
  The primary efficacy outcome is the difference of the change in the opaqueness of the carious lesion on the x-ray picture from Day 0 to Day 365 between test and control group.

SECONDARY OUTCOMES:
Additional benefit of a second Curodont Repair application | Day 720
  The secondary efficacy outcome is the difference of the change in the opaqueness of the carious lesion on the x-ray picture from Day 360 to Day 720 between test and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Seifert, Med. dent., Principal Investigator — Zahnheilkunde Seifert Gmbh
Locations (1):
- Zahnheilkunde Seifert Gmbh, Sirnach, Thurgau, Switzerland

REFERENCES:
- [Background] Brunton PA, Davies RP, Burke JL, Smith A, Aggeli A, Brookes SJ, Kirkham J. Treatment of early caries lesions using biomimetic self-assembling peptides--a clinical safety trial. Br Dent J. 2013 Aug;215(4):E6. doi: 10.1038/sj.bdj.2013.741. PMID 23969679